CLINICAL TRIAL: NCT01492166
Title: A Multi-center, Prospective, Non-interventional Evaluation of Efficacy, Safety and Convenience of Mixtard® 30 NovoLet® as Monotherapy, or in Combination With Oral Hypoglycaemic Agent ( OHA ), in Treatment of Subjects With Type 2 Diabetes in Routine Clinical Practice
Brief Title: Observational Study on Efficacy, Safety and Convenience of Using Mixtard® 30 NovoLet® Alone or Combined With OHA in Treatment of Type 2 Diabetes in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NOPEN3-1890
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — biphasic human insulin 30

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Novolet®
  Interventions: Drug: biphasic human insulin 30

INTERVENTIONS:
Drug: biphasic human insulin 30 — Dose and timing of dose for each subject was at the discretion of the attending physicians based on current clinical practice guidelines

SUMMARY:
This study is conducted in Asia. The aim of this study is to assess the efficacy, safety and convenience of the use of Mixtard® 30 NovoLet® used alone or combined with oral hypoglycaemic agent (OHA) in the management of type 2 diabetes mellitus in an out-patient setting.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Not adequately controlled on their current therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with type 2 diabetes not achieving adequate control and being prescribed Mixtard® 30 Novolet® either as a single treatment or in combination with oral hypoglycaemic agents (OHAs).
Sampling Method: Probability Sample
Enrollment: 1935 (Actual)
Dates: Start 2006-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in fasting blood glucose (FBG)
Change in 2-hour post prandial blood glucose
Change in HbA1c (glycosylated haemoglobin)
Change in prandial glucose increment (PGI)

SECONDARY OUTCOMES:
Frequency of minor and major hypoglycaemia
Occurrence of Adverse Drug Reactions (ADR)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Jakarta, Indonesia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com